CLINICAL TRIAL: NCT02623361
Title: A Prospective Analysis of Preoperative Fascia Iliaca Block for Hip Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FICB for hip athroscopy
Record Dates: First submitted 2015-12-01; First posted 2015-12-07 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Muscle Weakness | Patient; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham (Placebo Comparator)
  Interventions: Drug: Sham Block
- Fascia Iliaca Compartment Block (Active Comparator)
  Interventions: Drug: Peripheral Nerve Block

INTERVENTIONS:
Drug: Peripheral Nerve Block — Regional Anesthesia by Local Anesthetic Injection
  Arms: Fascia Iliaca Compartment Block
Drug: Sham Block — Sham Block by saline injection
  Arms: Sham

SUMMARY:
Patients undergoing arthroscopic hip surgery have been shown to have significant post-operative pain that may delay discharge, recovery, and early mobilisation. A pre-operative regional anesthesia technique, the fascia iliaca block may be an effective method for acute post-operative analgesia.

This is a prospective, randomized controlled study of the preoperative fascia iliaca block for patients undergoing hip arthroscopy.

The enrolled patients will be randomized to receive either a fascia iliaca block with the local anesthetic ropivacaine or to have a sham block. All patients will receive a general anesthetic for the hip arthroscopy.

DETAILED DESCRIPTION:
Arthroscopic hip surgery is used to diagnose and treat interior joint pathology. Although minimally invasive in nature, patients have considerable amount of pain postoperatively, leading to prolonged recovery room stay and increased opiate requirements. The investigators performed a retrospective chart review in patients who underwent hip arthroscopy at the UCSF Orthopedic Institute. 89% of the patients had pain immediate after surgery requiring opioid therapy. Regional anesthesia has previously been shown to reduce discomfort after hip arthroscopy. However, there is currently no safe, well-established ultrasound guided regional anesthesia technique for arthroscopic hip surgery. The fascia iliaca block has shown to decrease acute pain related with hip fractures, as well as pain related with knee arthroplasty. The ultrasound guided fascia iliaca block is easy to perform and has an excellent safety record. The investigators believe that the ultrasound guided fascia iliaca block improves pain control in patients undergoing arthroscopic hip surgery.

Patients will receive a sham block group or a fascia iliaca block, performed in the preoperative area.

Pain scores and measurement of quadriceps strength will be assessed preoperatively and postoperatively. The patient will receive a pain diary consisting of pain scores, pain medication consumption, and a brief pain inventory. Within 48 hours postoperatively, an anesthesiologist will call the patient and review the patient's pain scores, pain medication consumption and brief pain inventory.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* American Society of Anesthesia physical classification I - III, scheduled for arthroscopic hip surgery

Exclusion Criteria:

* Age younger than 18 years old
* Non-English speaking
* Contraindicated for regional nerve block (such as, but not limited to: coagulopathy, infection at site, allergy to local anesthetic)
* Preexisting neurologic deficits of operative limb
* Need for postoperative nerve function test
* Inability to consent due to cognitive dysfunction
* Chronic pain
* Patient refusal.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Behrends, MD, Principal Investigator — University of California
Locations (1):
- Orthopedic Institute, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FICB: Peripheral Nerve Block: Regional Anesthesia by Local Anesthetic Injection
Period: Overall Study
Arm/Group | Sham | FICB
Started | 40 | 40
Completed | 40 | 38
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | FICB | Total
Number analyzed (Participants) | 40 | 38 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (9) | 35 (11) | 34 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 17 | 23 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40 | 38 | 78

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Score
Description: highest reported numeric score 0-10 in Post Anesthesia Care Unit (PACU) (primary endpoint) The NRS score is used to rate pain from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: within one hour after surgery
Population: Exclusion criteria for enrollment included age younger than 18 years, contraindications for regional anesthesia, pre-existing neurologic deficits of the lower extremity, and a history of chronic pain requiring chronic opioid medication.
Measure: Mean (Standard Deviation); unit: units on the numeric rating scale (0-10)
Arm/Group | Sham | FICB
Number analyzed (Participants) | 40 | 38
units on the numeric rating scale (0-10) | 7 (2) | 6 (2)

2. Secondary Outcome: Leg Strength at Discharge From Ambulatory Center, Surgical Leg
Description: measurement of quadriceps strength (Force) using a dynamometer
Time Frame: 2 hours after surgery
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Sham | FICB
Number analyzed (Participants) | 40 | 38
Newton | 139 (99) | 41 (61)

3. Secondary Outcome: Patient Satisfaction
Description: patient questionaire, patients are contacted 48 h after surgery
  patient satisfaction is assessed using a questionnaire, applying a scale from 0 to 10, with 0 indicating "not satisfied at all" and 10 indicating "very satisfied"
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on the numeric rating scale (0-10)
Arm/Group | Sham | FICB
Number analyzed (Participants) | 37 | 38
units on the numeric rating scale (0-10) | 10 (0) | 10 (1)

ADVERSE EVENTS:
Arm/Group | Sham | FICB
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 0/40 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No